CLINICAL TRIAL: NCT00586547
Title: A Phase I Trial Evaluating The Use of RFT5-dgA to Deplete Alloreactive Cells PriorTo Haploidentical Stem Cell Transplantation
Brief Title: Evaluating the Use of RFT5-dgA to Deplete Alloreactive Cells Prior to Haploidentical Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of Texas, Southwestern Medical Center at Dallas (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Dist Serv Prof, Center for Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-9033; NCT00622297 (obsolete NCT alias)
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Leukemia; Cancer
Keywords: Haploidentical; Stem Cell Transplant; Graft-Versus-Host disease
MeSH Terms: conditions — Leukemia; Neoplasms; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): After patients have completed preparation to receive cells, they will be treated at one of five dose levels.
  Interventions: Biological: T-Cell Infusion Dose Level -1; Biological: T-Cell Infusion Dose Level 1; Biological: T-Cell Infusion Dose Level 2; Biological: T-Cell Infusion Dose Level 3; Biological: T-Cell Infusion- Dose Level 4

INTERVENTIONS:
Biological: T-Cell Infusion Dose Level -1 — (1 x 10^3 T cells/Kg)
Biological: T-Cell Infusion Dose Level 1 — (1 x 10^4 T cells/Kg)
Biological: T-Cell Infusion Dose Level 2 — (1 x 10^5 T cells/Kg)
Biological: T-Cell Infusion Dose Level 3 — (1 x 10^6 T cells/Kg)
Biological: T-Cell Infusion- Dose Level 4 — (5 x 10^6 T cells/Kg)

SUMMARY:
This study is designed to determine the number of donor lymphocytes that can be given to recipients of haploidentical stem cell transplants after depletion of recipient-reactive T lymphocytes by ex-vivo treatment with a fixed dose of RFT5-dgA immunotoxin, and will result in a rate of Grade III/IV GVHD of < / = 25%, to analyze immune reconstitution in these patients, and to measure their overall and disease free survival, at 100 days and at 1 year.

DETAILED DESCRIPTION:
Patients will receive cytosine arabinoside (3g/m^2) IV every 12 hours for 6 doses starting at 1400 hours on day -8. Cyclophosphamide (45mg/kg) will be given on Day -7 and Day -6. MESNA (45mg/kg, divided into 5 doses) will be administered 15 minutes prior to each dose of cyclophosphamide and 3, 6, 9 and12 hours after each dose of cyclophosphamide. Campath 1H IV will be given on Days -3, -2 and -1. TBI, total dose 14.0 Gy will be delivered in 8 fractions of 1.75 Gy in two fractions per day beginning Day -4. The dose rate will be 10cGy/min.

Approximately thirty days following transplantation (day +30), the cryopreserved T cells will be thawed and infused through a catheter line with normal saline.

This study will begin with a dose of T cells known not to cause GvHD even in haploidentical recipients, even when the T cells administered have not first been allodepleted. A subset of patients who achieved engraftment will be included in the dose escalation study of allodepleted T-cells treated with RFT5-dgA. A continual reassessment method based on a logistic dose-response curve with cohorts of size 2 will be employed to determine the MTD. Cohorts of size 2 will be accrued beginning at dose level 1 and the dose-response curve is estimated after toxicity outcome is observed to determine the recommended dose level for the next patient cohort. Each and every patient will receive up to five additional injections of T cells at the same dose, at monthly intervals, provided there is no evidence of grade 2 or higher GVHD, until total T cell numbers are > 1000/ul

Patients will be entered starting at level 1, according to the following doses:

Dose level -1 (1 x 10^3 T cells/Kg); Dose level 1 (1 x 10^4 T cells/Kg); Dose level 2 (1 x 10^5 T cells/Kg); Dose level 3 (1 x 10^6 T cells/Kg); Dose level 4 (5 x 10^6 T cells/Kg).

ELIGIBILITY:
Inclusion Criteria:

* ALL or high grade NHL that is Stage III or IV and has relapsed or is considered to be primary refractory disease.
* Myelodysplastic syndrome.
* AML after first relapse or with primary refractory disease.
* CML hemophagocytic lymphohistiocytosis (HLH)
* Familial hemophagocytic lymphohistiocytosis (FLH)
* Viral-associated hemophagocytic syndrome (VAHS)
* X-linked lymphoproliferative disease (XLP)
* Patients with Severe chronic active Epstein Barr virus infection (SCAEBV) with predilection for T- or NK-cell malignancy
* Lack of suitable conventional donor (i.e. 5/6 or 6/6 related or 5/6 or 6/6 unrelated donor) or presence of a rapidly progressive disease not permitting time to identify an unrelated donor.
* Donor cells should be collected and frozen before conditioning starts.

Exclusion Criteria:

* Patients with a life expectancy (< or = to 6 weeks) limited by diseases other than leukemia.
* Patients with symptomatic cardiac disease, or evidence of significant cardiac disease by echocardiogram (i.e. shortening fraction < 25%)
* Patients with severe renal disease (i.e. creatinine clearance less than 40cc/1.73m2)
* Patients with pre-existing severe restrictive pulmonary disease (FVC less than 40% of predicted)
* Patients with severe hepatic disease (direct bilirubin greater than 3ug/dl or SGPT greater than 500ug/dl)
* Patients with severe personality disorder or mental illness that would preclude compliance with the study
* Patients with a severe infection that on evaluation by the Principal Investigator precluded ablative chemotherapy or successful transplantation
* Patients with documented HIV positivity

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2000-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Determining the number of donor lymphocytes given to recipients of haploidentical stem cell transplants after depletion of recipient-reactive T lymphocytes by ex-vivo treatment with a fixed dose of RFT5-dgA immunotoxin. | 100

SECONDARY OUTCOMES:
To measure their overall and disease free survival. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Brenner, MB, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Methodist Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas